CLINICAL TRIAL: NCT01497353
Title: Is the Placental Transfusion Volume Influenced by the Position of the New Born at Birth?
Brief Title: Placental Transfusion and Cord Clamping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Salud Materno Infantil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: funda04
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Placental Transfusion
Keywords: Cord clamping; newborn; Skin contact; Placental transfusion; Delivery room
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Position at introitus level (Active Comparator): The newborn will be held by the neonatologist at the level of the introitus, the cord will be clamped at 2 minutes after birth. New weigh will be obtained after that.
  Interventions: Procedure: Position at introitus level
- Position at Maternal Abdomen (Experimental): The newborn will be placed on the abdomen and of the mother immediately after the first weigh measurement. The cord will be clamped at 2 minutes after birth .
  Interventions: Procedure: position at Maternal Abdomen

INTERVENTIONS:
Procedure: Position at introitus level — After birth: Weigh at 10 + 2 sec then Held the baby at the level of introitus and Cord clamping will be performed at 120 sec then another Weigh will be obtained after clamping
  Arms: Position at introitus level
Procedure: position at Maternal Abdomen — After birth: Weight at 10 + 2 sec then the baby will be placed at maternal abdomen and Cord clamping will be performed at 120 sec and new Weigh will be obtained after clamping
  Arms: Position at Maternal Abdomen

SUMMARY:
To compare the evolution of the infant's weight before delayed cord clamping (2 minutes after birth) as an indirect measure of the volume of placental transfusion in a group of healthy and fullterm newborns, placed at the level of the introitus versus another group placed on the abdomen of the mother.

DETAILED DESCRIPTION:
No inferiority, Randomized controlled trial not blind, Multicenter. Informed consent will be obtained during pregnancy or admittance and previous to birth.

Hypothesis: Placing the infant on the maternal abdomen without cord clamping during the first 2 minutes after birth does not change significantly the transfusion volume as compared to infants whose cord is clamped after 2 minutes but who are placed at the level of the introitus

Term newborns by vaginal delivery and without complications will be included. Study subjects will be assigned to two groups, both with delayed clamping,according to a sequence of random numbers generated by computer. The assignment will be done through opaque, sealed, easy opening envelopes, opening the envelope at the moment the mother enters the delivery room. Both parents and obstetric group will be then informed about which group the infant will be assigned to.

In both groups: The newborn will be immediately placed on a scale, previously set at the level of the maternal introitus to record his/her weight.

Group 1: Clamping at level of introitus: The infant will be held by the neonatologist at introitus level,immediately after the initial weight Group 2: Clamping on Maternal Abdomen: The newborn will be placed on the abdomen of the mother immediately after the first weight measurement.

In both groups:A plastic clamp will be put at approximately 1cm from the cutaneous insertion of the umbilical cord at 120 seconds after birth and then a new Weight will be obtained after clamping.

Weight differences will be evaluated when positioning the infant at the level of the introitus or on the maternal abdominal-thoracic level (at or over placental level).

ELIGIBILITY:
Inclusion Criteria:

* Term newborns
* vigorous born by vaginal delivery
* informed consent Signed.

Exclusion Criteria:

* History of Placenta previa,
* postpartum hemorrhage background,
* Multiple gestation.
* Background of IUGR prenatally diagnosed.
* Major congenital malformations diagnosed previous to delivery.
* Maternal diseases such as: eclampsia, Rh incompatibility, congestive cardiac failure.
* Extraction of blood sample for bank of umbilical cord stem cells.

Elimination criteria:

* Need for immediate assistance of the newborn,
* Birth weight less than 2500 g,
* Nuchal cord wrapped too tight,
* Major congenital malformations not diagnosed during prenatal period,
* Delivery surgically finished Short umbilical cord which might prevent placing the infant in the assigned place .

Max Age: 2 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Compare infant's birth weight before delayed cord clamping as an indirect measure of the volume of placental transfusion in a group of healthy fullterm newborns placed at the level of the introitus versus at the the mother's abdomen. | inmediately after birth until 2 minutes after birth
  Every elegible and randomiced newborn will be Immediately after birth placed on a scale at the level of the introitus, and the infant's weight will be recorded at 10± 2 sec.
  Group 1: The infant will be held by the neonatologist at introitus level. The cord will be clamped at 120 seconds after birth.
  Group 2: The newborn will be placed on the abdomen of the mother immediately after the first weight measurement. The cord will be clamped at 120 seconds after birth.
  Both groups will be weigth after the cord clamping.

SECONDARY OUTCOMES:
To compare venous hematocrit and bilirubin values between the 2 groups. | 36-48 hs
  venous hematocrit and bilirubin will be taken together with the sample taken for the mandatory neonatal screening.

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Vain, MD, Principal Investigator — Fundasamin
Locations (3):
- Argentina (3):
  - Hospital Materno Infantil de San Isidro Dr. C. Gianantonio, San Isidro, Buenos Aires
  - Sanatorio de la Trinidad Palermo, Buenos Aires, Buenos Aires F.D.
  - Instituto de Meternidad y ginecología Nuestra señora de las Mercedes, San Miguel de Tucumán, Tucumán Province

REFERENCES:
- [Background] Fonseca D. Importancia del aporte de sangre placentaria al niño recién nacido. Su medida por medio del registro ponderal continuo.Arch. Pediatr.Uruguay 1962; 7: 444
- [Result] Rabe H, Reynolds G, Diaz-Rossello J. A systematic review and meta-analysis of a brief delay in clamping the umbilical cord of preterm infants. Neonatology. 2008;93(2):138-44. doi: 10.1159/000108764. Epub 2007 Sep 21. PMID 17890882
- [Result] Diaz-Rossello JL. A difficult ethics issue. Lancet. 2004 Nov 13-19;364(9447):1751-2; author reply 1752. doi: 10.1016/S0140-6736(04)17385-6. No abstract available. PMID 15541437
- [Result] Ceriani Cernadas JM, Carroli G, Pellegrini L, Otano L, Ferreira M, Ricci C, Casas O, Giordano D, Lardizabal J. The effect of timing of cord clamping on neonatal venous hematocrit values and clinical outcome at term: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):e779-86. doi: 10.1542/peds.2005-1156. Epub 2006 Mar 27. PMID 16567393
- [Result] McDonald SJ, Middleton P. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004074. doi: 10.1002/14651858.CD004074.pub2. PMID 18425897
- [Result] Chaparro CM, Neufeld LM, Tena Alavez G, Eguia-Liz Cedillo R, Dewey KG. Effect of timing of umbilical cord clamping on iron status in Mexican infants: a randomised controlled trial. Lancet. 2006 Jun 17;367(9527):1997-2004. doi: 10.1016/S0140-6736(06)68889-2. PMID 16782490
- [Result] Lind J. Physiological adaptation to the placental transfusion: the eleventh blackader lecture. Can Med Assoc J. 1965 Nov 20;93(21):1091-100. No abstract available. PMID 5321023
- [Result] Hutton EK, Hassan ES. Late vs early clamping of the umbilical cord in full-term neonates: systematic review and meta-analysis of controlled trials. JAMA. 2007 Mar 21;297(11):1241-52. doi: 10.1001/jama.297.11.1241. PMID 17374818
- [Result] Yao AC, Lind J. Placental transfusion. Am J Dis Child. 1974 Jan;127(1):128-41. doi: 10.1001/archpedi.1974.02110200130021. No abstract available. PMID 4588934
- [Result] van Rheenen PF, Brabin BJ. Effect of timing of cord clamping on neonatal venous hematocrit values and clinical outcome at term: a randomized, controlled trial. Pediatrics. 2006 Sep;118(3):1317-8; author reply 1318-9. doi: 10.1542/peds.2006-1053. No abstract available. PMID 16951036
- [Result] Moore ER, Anderson GC, Bergman N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003519. doi: 10.1002/14651858.CD003519.pub2. PMID 17636727
- [Result] Yao AC, Hirvensalo M, Lind J. Placental transfusion-rate and uterine contraction. Lancet. 1968 Feb 24;1(7539):380-3. doi: 10.1016/s0140-6736(68)91352-4. No abstract available. PMID 4169972
- [Result] Yao AC, Moinian M, Lind J. Distribution of blood between infant and placenta after birth. Lancet. 1969 Oct 25;2(7626):871-3. doi: 10.1016/s0140-6736(69)92328-9. No abstract available. PMID 4186454
- [Result] Farrar D, Airey R, Law GR, Tuffnell D, Cattle B, Duley L. Measuring placental transfusion for term births: weighing babies with cord intact. BJOG. 2011 Jan;118(1):70-5. doi: 10.1111/j.1471-0528.2010.02781.x. Epub 2010 Nov 18. PMID 21083868
- [Derived] Vain NE, Satragno DS, Gorenstein AN, Gordillo JE, Berazategui JP, Alda MG, Prudent LM. Effect of gravity on volume of placental transfusion: a multicentre, randomised, non-inferiority trial. Lancet. 2014 Jul 19;384(9939):235-40. doi: 10.1016/S0140-6736(14)60197-5. Epub 2014 Apr 17. PMID 24746755